CLINICAL TRIAL: NCT02777437
Title: Laparoscopic Surgery VS Laparoscopic Surgery + Neoadjuvant Chemotherapy for T4 Tumor of the Colon Cancer: A Prospective, Multi-Center, Randomized, Open-Label, Parallel Group Clinical Trial
Brief Title: Laparoscopic Surgery VS Laparoscopic Surgery + Neoadjuvant Chemotherapy for T4 Tumor of the Colon Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Zhejiang University (Other); Tongji University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FuDanLapT4
Record Dates: First submitted 2016-05-02; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; Laparoscopic Surgery; Neoadjuvant chemotherapy; T4
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic surgery (No Intervention): Patients with T4 colon cancer receive laparoscopic surgery only.
- Neoadjuvantive chemotherapy + Laparoscopic surgery (Experimental): Patients with T4 colon cancer receive neoadjuvantive chemotherapy and laparoscopic surgery.
  Interventions: Drug: XELOX or FOLFOX chemotherapy

INTERVENTIONS:
Drug: XELOX or FOLFOX chemotherapy — 4 cycles of XELOX or FOLFOX neoadjuvant chemotherapy before surgery
  Other Names: Xeloda+ OXA or OXA+ 5-FU
  Arms: Neoadjuvantive chemotherapy + Laparoscopic surgery

SUMMARY:
Primary Outcome Measures: Disease free survival

Secondary Outcome Measures:

Overall survival

Adverse events (Mortality, morbidity)

The proportion of completion of Laparoscopic Surgery

Estimated Enrollment: Oct, 2016

Study Start Date: Oct, 2016

Estimated Study Completion Date: Oct, 2019

Estimated Primary Completion Date: Oct, 2021

Groups/Cohorts

1. Laparoscopic surgery for T4 colon cancers
2. Neoadjuvantive chemotherapy + Laparoscopic surgery for T4 colon cancers

DETAILED DESCRIPTION:
Investigators' previous studies indicated that laparoscopic surgery is feasible in T4 colon cancers with comparable clinical and oncologic outcomes. Laparoscopy may be considered as an alternative approach for T4 colon cancers with the advantage of faster recovery. The survival outcome of T4 colon cancers still dismays clinicians and patients. Preoperative chemotherapy is an attractive concept for locally advanced colon cancer. Optimal systemic therapy at the earliest possible opportunity may be more effective at eradicating distant metastases than the same treatment given after the delay and immunological stress of surgery. Besides, the shrinkage of primary tumor before surgery may reduce the risk of incomplete surgical excision and the risk of shedding of tumor cells during surgery. The aim of the present study is to compare the short-and long-term survival outcomes between laparoscopic surgery alone and laparoscopic surgery with 4 cycles of neoadjuvant chemotherapy for T4 colon cancer as well as the mortality and the morbidity.

The number of patients, which needs to get power of 80%, is 1960. The average numbers of patients needs to reach approximately 200, and that of surgical centers needs to reach 10.

Arrangements in the preoperative, intraoperative and postoperative period will be in complete accordance with the usual care of the center.

The baseline demographics and conditions as well as the perioperative items and the postoperative occurrences will be recorded through a prior designed e-questionnaire.

Globally,the disease free survival rate (chemotherapy and surgery), mortality (chemotherapy and surgery), the morbidity (chemotherapy and surgery) and the proportion of completion of laparoscopic surgery of the two surgical strategies will be analized and compared.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Histologically confirmed diagnosis of colon carcinoma
* CT or MRI verified as T4 colon cancer without involvement of other organs.
* Without multiple lesions other than carcinoma in situ
* Tumor size < 8 cm
* No bowel obstruction
* Sufficient organ function
* No history of gastrointestinal surgery
* 18 years of age or older
* Performance Status (ECOG) 0, 1 or 2, life expectancy > 12 weeks
* Operable patients
* Completion of neoadjuvant systemic chemotherapy

Exclusion Criteria:

* Women who are pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding
* No intention to finish neoadjuvantive systemic therapy
* Unstable or uncompensated respiratory or cardiac disease
* Serious active infections
* Hypersensitivity to capecitabine/fluorouracil or oxaliplatin
* Stomatitis or ulceration in the mouth or gastrointestinal tract
* Severe diarrhea
* Peripheral sensory neuropathy with functional impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3-year
  calculated from the date of surgery to the date of recurrence

SECONDARY OUTCOMES:
Overall survival | 3-year
  calculated from the date of diagnosis to the date of death from any cause
Adverse events (mortality and morbidity) | 3-month
  Number of participants with treatment-related adverse events assessed by CTCAE v4.0
The proportion of completion of laparoscopic surgery | 1-month
  The number of completion of laparoscopic surgery/the number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Xinxiang Li, MD,PhD, Principal Investigator — Fudan University